CLINICAL TRIAL: NCT07034872
Title: Effect of Multidimensional Trunk-Focused Exercise Training on Postural Control, Gait, and Activity in Children With Cerebral Palsy
Brief Title: Effect of Multidimensional Trunk Training in Children With Cerebral Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Irem Nur Sener, Doctorate Student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUC2025/105
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Palsy (CP)
Keywords: postural control; activity; gait; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group will receive two face-to-face physiotherapy sessions and one asynchronous video-based exercise training session per week for eight weeks. In addition to conventional therapy, this group will undergo a trunk-focused exercise program for the same duration.
  Interventions: Other: Intervention Group
- Control Group (Active Comparator): Participants in the control group will receive two face-to-face physiotherapy sessions and one asynchronous video-based conventional therapy session per week for eight weeks.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Control Group — Participants in the control group will receive two face-to-face physiotherapy sessions and one asynchronous video-based exercise training session per week for eight weeks. Following the baseline assessments, a conventional exercise program will be individually planned by the physiotherapist for each child. Each 60-minute session will include strengthening exercises for upper and lower extremity muscles, active and passive stretching exercises for spastic muscles, static and dynamic balance training in standing, and gait exercises.
  Arms: Control Group
Other: Intervention Group — Following baseline assessments, a personalized 60-minute exercise program will be developed by the physiotherapist for each child in the intervention group, consisting of two face-to-face sessions and one asynchronous video-based session per week for eight weeks. Each session will include 30 minutes of multidimensional trunk-focused exercises-such as static and dynamic trunk control (e.g., reaching, rotational movements), scapular and pelvic mobilizations, isolated muscle training, proprioceptive activities, and core strengthening-followed by 30 minutes of conventional therapy, including upper and lower extremity strengthening, stretching for spastic muscles, balance training in standing, and gait exercises.
  Arms: Intervention Group

SUMMARY:
This study investigates the effects of a personalized, multidimensional trunk-focused exercise program combined with conventional rehabilitation on postural control, gait, selective motor control, spasticity, activity participation, and quality of life in children with spastic cerebral palsy. Participants will be randomly assigned to an intervention group receiving trunk-focused exercises plus conventional therapy or a control group receiving only conventional therapy over an eight-week period with thrice-weekly sessions (two face-to-face, one home-based via video guidance). The study also incorporates caregiver-supported home exercises facilitated by a web-based platform and mobile application to enhance adherence and sustainability. Outcomes will be assessed pre- and post-intervention to evaluate the program's efficacy in improving motor function and daily activity engagement.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is defined as a chronic condition characterized by non-progressive disorders that occur in early childhood and affect motor development, leading to functional limitations. Among the different types of CP, spastic CP is the most common. In children with spastic CP, impairments in the development of balance and protective reactions, associated reaction patterns, and stereotypical movement patterns form the basis of postural control deficits. Achieving trunk control during early childhood is considered a crucial indicator for future ambulation. It is known that age three is a critical milestone in the motor development of children with CP, and approximately one in three children cannot attain adequate trunk control for stable and independent sitting by this age. A moderate correlation has been reported between trunk control, balance parameters, and gait capacity in children with spastic CP.

Evaluating the clinical characteristics of impaired postural control in children with CP and applying appropriate rehabilitation methods is of great importance for promoting independence in activities of daily living. In CP rehabilitation, interventions aiming to improve postural control have shown moderate-quality evidence regarding the effectiveness of trunk-focused training. However, the absence of standardized protocols for such interventions remains a significant limitation in tailoring therapies to individual needs.

This study aims to contribute to the literature by investigating the potential effects of a personalized, multidimensional, trunk-focused exercise program implemented in addition to conventional rehabilitation on postural control development (including static and dynamic trunk control, standing balance, and gait), selective motor control, posture, spasticity level, activity and participation levels, and quality of life in children with spastic CP. Furthermore, the project aims to complement face-to-face therapies with home-based exercises guided by caregivers using individualized exercise prescriptions delivered through a web-based platform and mobile application. This approach is expected to enhance caregiver knowledge and competence, ensure regular exercise adherence, and support the sustainability of the therapeutic process at home.

Children with spastic cerebral palsy who meet the inclusion criteria will be evaluated in terms of trunk control, balance, posture, selective control of upper and lower extremities, spasticity, gait, activity and participation levels, and quality of life, and will be randomly assigned into two groups. The study will last for eight weeks, during which all participants will receive therapy three times per week: two face-to-face sessions with a physiotherapist and one home-based session using asynchronous video-guided exercises delivered via a web-based platform and/or mobile application, under caregiver supervision. During each session over the eight-week intervention period, the study group will receive 30 minutes of a multidimensional trunk-focused exercise program in addition to 30 minutes of conventional therapy, whereas the control group will receive 60 minutes of conventional therapy. At the end of the eighth week, all initial assessments will be repeated for both groups.

The study aims to demonstrate the effects of a personalized multidimensional trunk-focused exercise training program on postural control, gait, and activity levels in adolescents with spastic-type cerebral palsy. Furthermore, the sustainability of the therapeutic process will be supported through the home-based implementation of these exercises under caregiver supervision, facilitated by the web-based system and mobile application TeleRehab4Kids.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with spastic type cerebral palsy
* Aged between 9 and 18 years
* Classified as levels 1, 2, or 3 according to the Gross Motor Function Classification System (GMFCS)

Exclusion Criteria:

* Having received Botox injections targeting the upper and lower extremities within the last 6 months
* Diagnosed with mental retardation
* Having visual and/or hearing impairments severe enough to affect participation in treatment
* Lack of internet access at home and not possessing digital devices such as a smartphone, tablet, or computer
* Having an additional neurological disorder diagnosis other than cerebral palsy

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2026-10-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Trunk Control Measurement Scale (TCMS) | Baseline and after 8 weeks
  The TCMS consists of two main subcomponents: static and dynamic sitting balance. The static sitting balance section evaluates static trunk control during upper and lower extremity movements and has been shown to be a valid and reliable tool in children with cerebral palsy (Heyrman et al., 2011). The dynamic sitting balance section is further divided into two subcategories: selective movement control and dynamic reaching. The selective movement control subcomponent assesses the pelvis's ability to perform selective movements in all three planes (flexion-extension, lateral flexion, and rotation) while seated on a support surface. The dynamic reaching subcomponent evaluates performance during reaching tasks. The scale consists of 15 items, with a total score ranging from 0 to 58, where higher scores indicate better trunk control.
Pediatric Balance Scale (PBS) | Baseline and after 8 weeks
  The Pediatric Balance Scale is an adaptation of the Berg Balance Scale, originally developed for adults, for use in children. It is a functional balance assessment tool consisting of 14 items that evaluate parameters such as sitting to standing, standing, transfers, stepping, and turning (Franjoine M.R. et al., 2003). The scale has been validated for use in children with cerebral palsy in Turkish populations (Erden A. et al., 2021).

SECONDARY OUTCOMES:
Selective Control of the Upper Extremity Scale (SCUES) | Baseline and after 8 weeks
  The SCUES is designed for professionals to assess and score selective motor control of the upper extremities. It is a practical and easy-to-administer tool, as it requires no equipment other than a video camera. The assessed joint movements of the upper extremity include shoulder (abduction/adduction), elbow (flexion/extension), forearm (supination/pronation), wrist (flexion/extension), and fingers/thumb (grasp/release). The Turkish version of the scale has been validated for reliability and validity (Yildiz A. et al., 2022).
Selective Control Assessment of the Lower Extremity (SCALE) | Baseline and after 8 weeks
  The SCALE is a valid and reliable assessment tool designed to evaluate selective voluntary motor control of the lower extremities by assessing the hip, knee, ankle, subtalar, and toe joints individually and bilaterally (Fowler E.G. et al., 2009). The administration time is approximately 15 minutes and can be conducted either in-person or through video recordings. The tool consists of three components: application instructions, scoring guidelines, and a score sheet. Specific testing positions are provided for each joint assessed. The patient is instructed to perform each movement over approximately 3 seconds, guided by a verbal tempo. Each joint is scored as follows: "Normal = 2 points," "Impaired = 1 point," and "Unable = 0 points." The Turkish version of the SCALE has been validated for use in children with cerebral palsy (Tunçdemir M. et al., 2020).
PostureScreen Mobile® | Baseline and after 8 weeks
  PostureScreen Mobile® is a valid and reliable mobile application developed to facilitate postural assessment in various environments. It is a posture analysis, body composition, and movement assessment software designed for use on iOS and Android devices via the device's camera (Moreira R. et al., 2020).
Modified Ashworth Scale (MAS) | Baseline and after 8 weeks
  The Modified Ashworth Scale will be used to assess the effect of increased muscle tone in the upper and lower extremity muscle groups on postural control. When a joint is passively moved within its normal range of motion, the resistance of the muscle to this passive movement indicates the degree of spasticity. Muscle tone is rated on a six-point ordinal scale: 0, 1, 1+, 2, 3, and 4. A score of 0 indicates no increase in muscle tone, while a score of 4 reflects rigidity in flexion and extension of the affected muscle (Numanoğlu Akbaş A., 2016).
Edinburgh Visual Gait Score (EVGS) | Baseline and after 8 weeks
  The Edinburgh Visual Gait Score is a 17-item scale designed to represent key characteristics of gait in children with cerebral palsy. It assesses the trunk, pelvis, hip, knee, ankle, and foot in the sagittal, coronal, and transverse planes. A three-point ordinal scale is used for scoring (Robinson L.W. et al., 2017).
Timed Up and Go Test (TUG) | Baseline and after 8 weeks
  The Timed Up and Go Test measures the time it takes for an individual to rise from a chair with armrests, walk 3 meters, turn around, walk back to the chair, and sit down again. The time is recorded from the moment the individual begins to stand up until they are seated again. Prior to testing, the movement is demonstrated to the child. The test is performed twice, and the faster time is recorded. Durations under 10 seconds are considered normal, whereas times exceeding 14 seconds are indicative of a high risk of falling (Carey H. et al., 2016).
Pediatric Evaluation of Disability Inventory (PEDI) | Baseline and after 8 weeks
  The PEDI is a valid and reliable clinical assessment tool used to evaluate the functional status of children with cerebral palsy. The assessment comprises three domains: functional skills, caregiver assistance, and modifications, making it a comprehensive evaluation instrument for healthcare professionals in pediatrics (Haley S.M. et al., 1991). A Turkish validity and reliability study has also been conducted (Erkin G. et al., 2007).
Pediatric Outcomes Data Collection Instrument (PODCI) | Baseline and after 8 weeks
  This tool assesses health-related quality of life, functional health status, and participation in daily living activities. Its Turkish version has been validated and shown to be reliable in children aged 2 to 18 years diagnosed with cerebral palsy (Scott K.S. et al., 2021; Keskin Dilbay N. et al., 2013).
Participation and Environment Measure for Children and Youth (PEM-CY) | Baseline and after 8 weeks
  The PEM-CY is one of the most widely used tools to reflect children's participation in life activities (Khetani M. et al., 2014). It is utilized for children with cerebral palsy. The Turkish version has been validated and found reliable for clinical use and research purposes to assess participation and environmental factors in both disabled and non-disabled children and youth (Kaya Kara O. et al., 2020). This scale is the first parent-report questionnaire to evaluate children's participation across three key life settings-home (10 activities), school (5 activities), and community (10 activities)-while also addressing environmental factors.

OTHER OUTCOMES:
Clinical Assessment Form | Baseline
  Before conducting detailed evaluations, demographic and clinical data will be collected for each participant and documented in the patient and family records, including:
  Age (years), Height (cm), Weight (kg), Body Mass Index (BMI), Sex, Prenatal-perinatal-postnatal history, current rehabilitation status, and duration, implementation of home exercise program, history and timing of any surgical interventions within the past year, administration and timing of Botulinum toxin-A injections within the last 6 months, use of assistive devices, medication usage

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No